CLINICAL TRIAL: NCT06700707
Title: Turkish Adaptation, Validity and Reliability Study
Brief Title: Turkish Adaptation, Validity and Reliability Study of the Athlete Disability Index Questionnaire
Acronym: ADI_Turkish
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gülay Aras Bayram, Associate professor, Medipol University
Other Study IDs: 20112024
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain; Disability; Athlete; Sport
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey using a questionnaire. — Permission was obtained from the original owner of the Athlete Disability Index Questionnaire (ADI) for the Turkish cultural adaptation, validity and reliability study.
  120 athletes, determined by the number of questions times the rule of 10, will be asked to fill out the ADI, Oswestry Disability Index (ODI), and Roland-Morris Disability (RMDQ) questionnaires and 60 athletes will be asked to fill out the ADI questionnaire again 7 days later for test-retest reliability.

SUMMARY:
This survey study aims to analyze the cultural adaptation, validity, and reliability of a scale originally in English and currently being translated into Turkish, which allows athletes with low back pain to assess their functional disabilities in sports and exercise activities as well as their disabilities in daily living activities. Athletes with low back pain will be asked to fill out 3 questionnaires.

DETAILED DESCRIPTION:
In the study, firstly, the translation of the Athlete Disability Index Questionnaire (ADI) into the target language, comparison of the two translated versions of the scale, back translation of the preliminary version, synthesis, pilot test of the pre-final version and psychometric test studies will be carried out by 3 independent translators and 2 linguists in 6 stages.

Then, 120 athletes with low back pain will be asked to fill out the ADI, Roland Morris Disability Questionnaire (RMDQ) and Oswestry Low Back Pain Disability Index (ODI). 7 days later, the ADI will be filled out again by 60 athletes.

After the surveys are completed, the structural validity of the scale will be tested, and reliability will be measured by performing test-retest reliability and internal consistency analyses.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain that has persisted for at least 6 weeks
* Pain that worsens with changes in posture, movement, or physical activity
* Elite athletes with a regular training/match schedule of more than 10 hours per week

Exclusion Criteria:

* Not knowing Turkish
* Acute inflammatory conditions
* Acute musculoskeletal trauma
* Long-term corticosteroid use

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male and female elite athletes from different sports with low back pain
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Athlete Disability Index Questionnaire (ADI) | 7 days
  The Athlete Disability Index Questionnaire (ADI) is a self-administered questionnaire to assess disability related to low back pain in athletes. The ADI measures athletes' functional disability in activities of daily living as well as their disability in sports and exercise activities. The ADI consists of 12 questions that include pain intensity, stretching exercises, strengthening/weight training exercises, sport-specific skills (technical skills), rotational waist movements/changing direction, fear of pain or re-injury, sitting, walking, recreational activities, sexual activity, sleep, and personal care (ability to put on socks and shoes, ability to go to the bathroom). Each question is scored from 0 to 3, with higher scores indicating a more severe condition.

SECONDARY OUTCOMES:
Oswestry Low Back Pain Disability Index (ODI) | 1 day
  Oswestry Low Back Pain Disability Index (ODI) is a Likert-type scale that questions pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sexual life, social life and traveling in 10 items. Each item is scored between 0-5 (0: normal, 5: maximum difficulty) and the total score is 50.
  In it's calculation; (Final score = [total score] / [(number of marked questions) x5] x 100) formula is used to convert it to a percentage system. A high percentage indicates that the level of disability perceived by the patient is also high. Turkish validity and reliability study has been conducted.
Roland Morris Disability Questionnaire (RMDQ) | 1 day
  Roland Morris Disability Questionnaire (RMDQ): This scale, which was developed by selecting 24 of the 136 items of the Disease Impact Profile, evaluates activity level, daily living activities, eating and sleeping. Yes is scored as 1, no is scored as 0, and a higher total score indicates worse functionality. A Turkish validity and reliability study was conducted by Küçükdeveci et al.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Aras Bayram, PhD, Principal Investigator — Medipol University
Locations (1):
- Gülay Aras Bayram, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zamani E, Kordi R, Nourian R, Noorian N, Memari AH, Shariati M. Low back pain functional disability in athletes; conceptualization and initial development of a questionnaire. Asian J Sports Med. 2014 Dec;5(4):e24281. doi: 10.5812/asjsm.24281. Epub 2014 Nov 10. PMID 25741417
- See also: Link to the original article of the ADI survey — https://pubmed.ncbi.nlm.nih.gov/25741417/